CLINICAL TRIAL: NCT07377253
Title: A Phase I Study to Investigate the Safety, Tolerability, and Pharmacokinetic Characteristics of Intravenous (IV) Administration of a Human Monoclonal Antibody Against Tick-borne Encephalitis Virus in Healthy Adults.
Brief Title: First-in-Human Study Testing a New Antibody Treatment for Tick-Borne Encephalitis in Healthy Volunteers.
Acronym: SVRI01
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Giuseppe Pantaleo (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Pantaleo, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SVRI01
Record Dates: First submitted 2025-11-18; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: The Tick-borne Encephalitis Virus (TBEV)
Keywords: Tick-borne encephalitis; Tick-borne encephalitis virus; Human antibody therapy; Healthy volunteers; Phase I clinical trial; Intravenous administration; Monoclonal antibody
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: Phase I, Dose escalation 3+3, Non randomized, Open Label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): TBE025 200 mg administered intravenously on Day 0
  Interventions: Drug: Human monoclonal antibody TBE025, intravenous infusion
- Cohort 2 (Experimental): TBE025 600 mg administered intravenously on Day 0
  Interventions: Drug: Human monoclonal antibody TBE025, intravenous infusion
- Cohort 3 (Experimental): TBE025 2000 mg administered intravenously on Day 0
  Interventions: Drug: Human monoclonal antibody TBE025, intravenous infusion

INTERVENTIONS:
Drug: Human monoclonal antibody TBE025, intravenous infusion — TBE025 is a recombinant, fully human monoclonal antibody (mAb). It is provided in single-use vials containing 20 mg/mL of protein in 5 mL of buffered solution consisting of 10 mM Histidine, 250 mM Trehalose, 10 mM Methionine, 0.05% Polysorbate 20 and water for injection, at pH 5.5. TBE025 is a clear to opalescent, colorless to brown liquid.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and pharmacokinetics of the investigational monoclonal antibody TBE025 when given intravenously to healthy adult volunteers aged 18 to 55.

The study aims to determine the recommended Phase II dose of TBE025 and to assess the incidence and severity of adverse events related to its administration.

There is no comparison group, as this is a single-arm, open-label study. Participants will receive a single intravenous infusion of TBE025 at one of three escalating dose levels, will be monitored for safety with regular clinical and laboratory assessments, and will provide blood samples for pharmacokinetic, anti-drug antibody, and neutralization testing.

DETAILED DESCRIPTION:
The tick-borne encephalitis virus (TBEV) is an infection spread by ticks that is becoming more common in Europe, including Switzerland. Currently, there is no specific treatment-care focuses on relieving symptoms. Vaccines exist, but few people get vaccinated, and sometimes the vaccine does not offer full protection. There is therefore a real need for new ways to prevent or treat this disease.

TBE025 is a fully human antibody taken from people who have recovered from TBEV. It can strongly block the virus. In lab studies with mice, TBE025 was able to protect against infection, both when given before exposure and soon after infection. It also appears to be safe, with no harmful effects on other tissues.

This first-in-human study (phase 1) will evaluate intravenous administration of TBE025 in healthy adult volunteers using a standard 3+3 dose-escalation design (200 mg, 600 mg, 2000 mg). Between 3 and 18 participants will be enrolled sequentially across three cohorts. The study is designed to establish the maximum tolerated dose and recommended Phase II dose, as well as to characterize the pharmacokinetics, immunogenicity, and neutralization capacity of TBE025.

Participants will be followed for safety, laboratory, and pharmacokinetic assessments over a three-month period. The study will provide the first clinical data on TBE025 in humans and will inform the design of subsequent efficacy trials in populations at risk of TBEV infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to <55 years
* Good general health (medical history, physical exam, normal labs)
* Written informed consent provided
* Ability to read and understand local language
* Contraception requirements : Women of childbearing potential: negative pregnancy test, surgically sterile, postmenopausal, or using highly effective contraception for 3 months post-infusion. Men: surgically sterile or using highly effective contraception (self or partner) and abstain from sperm donation for 3 months post-infusion.

Exclusion Criteria:

* BMI <19 or >30
* Infections: HIV, active hepatitis B (HBsAg), active hepatitis C
* Prior participation in investigational study within 30 days
* History of hypersensitivity to monoclonal antibodies
* Recent surgery or unresolved adverse events
* Active autoimmune disease requiring systemic treatment
* Recent use of immunosuppressive agents or immunoglobulins
* Immunodeficiency diagnosis
* Significant cardiovascular events within 6 months
* Live/attenuated vaccines within 28 days
* Major surgery within 28 days
* Pregnancy or breastfeeding
* Professional or private link with the research team
* Any condition judged by the investigator to interfere with safety or study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of TBE025 | Up to 84 days after the infusion
  Number and percentage of subjects experiencing AEs, SAEs, AEs related to investigational product at each dose level
Incidence and severity of adverse events (AEs) | Up to 84 days after the infusion
  Number and percentage of subjects experiencing AEs related to investigational product and the severity of the AEs at each dose level
Incidence and severity of Dose Limiting Toxicity (DLT) | Up to 21 days after the infusion.
  Number and percentage of participants experiencing DLTs at each dose level.

SECONDARY OUTCOMES:
Pharmacokinetic profile of TBE025 | up to 84 days after infusion
  Plasma concentration measured by ELISA for each participant at each dose level
Presence of anti-drug antibodies | Up to 84 days after infusion
  Antibodies against TBE025 measured by ELISA for each participant at each dose group

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Universitaire Hospitalier Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. Only de-identified subject-level data may be provided if requested, and only in accordance with participant informed consent and applicable laws.